CLINICAL TRIAL: NCT03600909
Title: A Phase II Trial of Hematopoietic Stem Cell Transplantation for the Treatment of Patients With Fanconi Anemia Lacking a Genotypically Identical Donor, Using a Risk-Adjusted Chemotherapy Only Cytoreduction With Busulfan, Cyclophosphamide and Fludarabine
Brief Title: A Study of the Effect of Blood Stem Cell Transplant After Chemotherapy Alone in Patients With Fanconi Anemia
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Accrual has been slow
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: Pediatric Brain Tumor Consortium (Network)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 17-498
Record Dates: First submitted 2018-07-17; First posted 2018-07-26 (Actual); Results first posted 2022-04-12 (Actual); Last update posted 2022-04-12 (Actual); Status verified 2021-04

CONDITIONS: Fanconi Anemia; Myelodysplastic Syndrome (MDS); Acute Myelogenous Leukemia (AML)
Keywords: Blood Stem Cell Transplant; busulfan; cyclophosphamide; fludarabine; 17-498
MeSH Terms: conditions — Fanconi Anemia; Myelodysplastic Syndromes; Leukemia, Myeloid, Acute | interventions — Busulfan; fludarabine; fludarabine phosphate; Cyclophosphamide; Antilymphocyte Serum; Granulocyte Colony-Stimulating Factor; Filgrastim

STUDY DESIGN:
Intervention Model Description: A three-arm phase II treatment protocol designed to examine engraftment, toxicity, graft-versus-host disease, and disease-free survival following a novel cytoreductive regimen including busulfan, cyclophosphamide and fludarabine and ATG
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: Yes

ARMS (3):
- Good Risk Patients (Experimental): Patients 18 years old or younger with marrow aplasia or single lineage cytopenias (Arm A) will be conditioned for transplantation with intravenous busulfan (busulfex®) (0.6-0.8 mg/Kg/dose q 12 hours x 4 doses), cyclophosphamide (10 mg/Kg/dose x 4 doses) and fludarabine (35mg/m2/day x 4 doses).
  Interventions: Drug: Busulfan; Drug: Fludarabine; Drug: Cyclophosphamide; Drug: Anti-Thymocyte Globulin (Rabbit); Device: The CliniMACS device; Drug: G-CSF
- Intermediate risk patients (Experimental): Patients 18 years old or younger with MDS or AML will be will be conditioned for transplantation with intravenous busulfan (busulfex®) (0.8-1.0mg/Kg/dose q 12 hours x 4 doses), cyclophosphamide (10 mg/Kg/dose x 4 doses) and fludarabine (35mg/m2/day x 4 doses).
  Interventions: Drug: Busulfan; Drug: Fludarabine; Drug: Cyclophosphamide; Drug: Anti-Thymocyte Globulin (Rabbit); Device: The CliniMACS device; Drug: G-CSF
- High risk patients (Experimental): Patients 19 years old or older with marrow aplasia or MDS or AML will be will be conditioned for transplantation with intravenous busulfan (busulfex®) (0.4mg/Kg/dose q 12 hours x 4 doses), cyclophosphamide (10 mg/Kg/dose x 4 doses) and fludarabine (35mg/m2/day x 4 doses).
  Interventions: Drug: Busulfan; Drug: Fludarabine; Drug: Cyclophosphamide; Drug: Anti-Thymocyte Globulin (Rabbit); Device: The CliniMACS device; Drug: G-CSF

INTERVENTIONS:
Drug: Busulfan — A standard dose of busulfan, associated with excellent outcomes in our previous trial will be used for young patients with marrow aplasia (arm A).
  A higher dose of busulfan will be used in younger patients with MDS and AML (arm B) to maximize disease control.
  A lower dose of busulfan will be used in older patients (arm C) to minimize toxicity.
  Other Names: busulfex®
Drug: Fludarabine — Arms A, B and C - Fludarabine will be given IV over 30 minutes daily for 4 days. The dose will be adjusted according to renal function according to Institutional guidelines.
  Other Names: FLUDARA®
Drug: Cyclophosphamide — Arms A, B and C - Cytoxan will be given as a 1-2 hour infusion for 4 days. The dose will be adjusted according to patients ideal body weight for obese patients.
  Other Names: Cytoxan®
Drug: Anti-Thymocyte Globulin (Rabbit) — Arms A, B and C - 4 doses will be given prior to transplant to promote engraftment
  Other Names: hymoglobulin®
Device: The CliniMACS device — The source of stem cells for all patients will be peripheral blood stem cells (PBSC) induced and mobilized by treatment of the donor with G-CSF for 4-6 days. T-cell depletion will be uniformly performed by positive CD34 selection with the use of the Miltenyi system (CliniMACS device)
Drug: G-CSF — All patients will also receive G-CSF post-transplant to foster engraftment.
  Other Names: Granulocyte colony-stimulating factor, filgrastim

SUMMARY:
The goal of this study is to see if the study therapy can decrease the chemotherapy-related side effects while maximizing the effectiveness of disease control. The physicians will also be studying the effect of removing T-cells from the donor"s stem cells before transplant. T-cells are a type of white blood cell that may help cause a serious side effect of transplant called Graft versus Host Disease (GVHD). The way it removes the T-cells from the donor stem cells is actually by selecting only the stem cells (called CD34 cells) by using a device called CliniMACS. This process is called CD34 selection. The CliniMACS® device is currently under the supervision of the FDA .

ELIGIBILITY:
Inclusion Criteria:

* Patients must have a diagnosis of Fanconi anemia (confirmed by mitomycin C or diepoxybutane [DEB] chromosomal breakage testing at a CLIA approved laboratory).

Patients must have one of the following hematologic diagnoses:

1. Severe Aplastic Anemia (SAA), with bone marrow cellularity of <25% OR Severe Isolated Single lineage Cytopenia

AND at least one of the following features:

1. Platelet count <20 x 10^9/L or platelet transfusion dependence*
2. ANC <1000 x 10^9/L
3. Hgb <8 gm/dl or red cell transfusion dependence*

2. Myelodysplastic Syndrome (MDS) (Appendix 1: MDS Classification)

MDS at any stage, based on either one of the following classifications:

* WHO Classification
* Refractory anemia and transfusion dependence*
* Any of other stages
* IPSS Classification
* Low risk (score 0) and transfusion dependence*
* Any other risk groups Score > 0.5 Note that patients with chromosome 1q cytogenetic abnormalities in the absence of morphologic dysplasia will not be considered to have MDS.

  3. Acute Myelogenous Leukemia Patients with acute leukemia are included in this trial untreated, in remission or with refractory or relapsed disease.

  * Transfusion dependence will be defined as greater than ONE transfusion of platelets or red blood cells in the last year prior to evaluation on protocol.

Donor

Donor choices will be determined by the investigators according to institutional criteria. Patients who will be enrolled on this protocol must have one of the following donor choices:

HLA-compatible unrelated volunteer donors Patients who do not have a related HLA-matched donor but have an unrelated donor who is either matched at all A, B, C and DRB1 (8/8) loci or who is mismatched at no more than 2/8 loci (A, B, C or DRB1) (6/8) as tested by DNA analysis (high resolution), will be eligible for entry on this protocol.

HLA-mismatched Related donors Patients who do not have a related or unrelated HLA-compatible donor must have a healthy family member who is at least HLA-haplotype identical to the recipient. First degree related donors must have a normal DEB test.

The donor must be healthy and willing and able to receive a 4-6 day course of G-CSF and undergo 1-3 daily leukaphereses, as per institutional guidelines.

Related and unrelated donors must be medically evaluated and fulfill the criteria for collection of PBSCs as per institutional guidelines.

Patients and donors may be of either gender or any ethnic background. Patients must have a Karnofsky adult, or Lansky pediatric performance scale status ≥ 70%.

Patients must have adequate physical function measured by :

1. Cardiac: asymptomatic or if symptomatic then 1) LVEF at rest must be ≥ 50% and must improve with exercise or 2) Shortening Fraction ≥ 29%
2. Hepatic: < 5 x ULN alanine transaminase (ALT) and < 2.0 mg/dl total serum bilirubin.
3. Renal: serum creatinine ≤1.5 mg/dl or if serum creatinine is outside the normal range, then CrCl > 50 ml/min/1.73 m^2
4. Pulmonary: asymptomatic or if symptomatic, DLCO > 50% of predicted (corrected for hemoglobin) Each patient must be willing to participate as a research subject and must sign an informed consent form. Parent or legal guardians of patients who are minors will sign the informed consent form. Assents will be obtained as per institutional guidelines.

Female patients and donors must not be pregnant or breastfeeding at the time of signing consent. Women must be willing to undergo a pregnancy test prior to transplant and avoid becoming pregnant while on study. Positive pregnancy test results will be reported to the parent(s) or guardian of minor participants, as required per institutional guidelines.

Exclusion Criteria:

Active CNS leukemia Female patients who are pregnant (positive serum or urine HCG) or breast-feeding. Women of childbearing age must avoid becoming pregnant while on study.

Active uncontrolled viral, bacterial or fungal infection Patient seropositive for HIV-I/II; HTLV -I/II

Min Age: 1 Month | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2018-05-15 (Actual); Primary Completion 2021-04-09 (Actual); Study Completion 2021-04-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Farid Boulad, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (3):
- United States (3):
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Fred Hutchinson Cancer Research Center, Seattle, Washington

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/mskcc/html/44.cfm

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Good Risk Patients | Intermediate Risk Patients | High Risk Patients
Started | 0 | 3 | 0
Completed | 0 | 0 | 0
Not Completed | 0 | 3 | 0
Not completed — Not treated | 0 | 3 | 0

BASELINE CHARACTERISTICS:
Population: Study closed due to slow accrual
Groups:
- Total: Total of all reporting groups
Arm/Group | Good Risk Patients | Intermediate Risk Patients | High Risk Patients | Total
Number analyzed (Participants) | 0 | 3 | 0 | 3
Age, Continuous [Median (Full Range); unit: years] |  | 18 [7 to 24] |  | 18 [7 to 24]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female |  | 2 |  | 2
  Male |  | 1 |  | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino |  | 0 |  | 0
  Not Hispanic or Latino |  | 3 |  | 3
  Unknown or Not Reported |  | 0 |  | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native |  | 0 |  | 0
  Asian |  | 2 |  | 2
  Native Hawaiian or Other Pacific Islander |  | 0 |  | 0
  Black or African American |  | 0 |  | 0
  White |  | 1 |  | 1
  More than one race |  | 0 |  | 0
  Unknown or Not Reported |  | 0 |  | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States |  | 3 |  | 3

OUTCOME MEASURES:

1. Primary Outcome: Graft Failure or Rejection
Description: Primary non-engraftment is diagnosed when the patient fails to achieve an ANC ≥500/µl at any time in the first 28 days post-transplant. If (1) after achievement of an ANC ≥500/mm^3, the ANC declines to <500/mm^3 for more than 3 consecutive days in the absence of relapse, or, (2) there is absence of donor cells in the marrow and/or blood as demonstrated by chimerism assay in the absence of relapse, a diagnosis of secondary graft failure is made. The patient is not evaluable for graft failure or rejection if recurrence of host MDS is detected concurrently.
Time Frame: 5 years
Population: Data were not collected. No participants received treatment and study terminated due to slow accrual
Arm/Group | Good Risk Patients | Intermediate Risk Patients | High Risk Patients
Number analyzed (Participants) | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Up to 1 year
Description: All-Cause Mortality, Serious, or Other (non-serious) Adverse Events were monitored/assessed in the "Intermediate Risk Patients" Arm/Group but none observed.
Arm/Group | Good Risk Patients | Intermediate Risk Patients | High Risk Patients
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/3 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/3 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/3 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-03-08): https://cdn.clinicaltrials.gov/large-docs/09/NCT03600909/Prot_SAP_000.pdf